CLINICAL TRIAL: NCT02276950
Title: HeAlth-data Register sTudies of Risk and Outcomes in Cardiac Surgery (HARTROCS)
Brief Title: HeAlth-data Register sTudies of Risk and Outcomes in Cardiac Surgery
Acronym: HARTROCS
Status: Active, not recruiting | Type: Observational
Sponsor: Ulrik Sartipy, MD, PhD (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Ulrik Sartipy, MD, PhD, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: HARTROCS
Record Dates: First submitted 2014-10-25; First posted 2014-10-28 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases; Kidney Diseases; Depression; Diabetes Mellitus
Keywords: Cardiac Surgery; Epidemiologic Methods; Blood Transfusions
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Diseases; Depression; Diabetes Mellitus | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Coronary artery bypass surgery — Primary isolated coronary artery bypass surgery with or without use of cardio-pulmonary bypass
  Other Names: CABG
Procedure: Heart valve surgery — Heart valve surgery, aortic valve replacement or other heart valve procedures

SUMMARY:
The overall project aim is to study risk and outcomes following cardiac surgery by cross-linking high-quality national Swedish health-data registers for population-based investigations of individual level clinically relevant patient data.

DETAILED DESCRIPTION:
The purpose of this research project is to study risks and outcomes in patients who underwent cardiac surgery. We aim to establish a fundament for the conduct of nationwide population-based studies by linking patient-level data from the Swedish Heart Surgery Register (SWEDEHEART), the National Patient Register, the Cause of Death Register, the National Diabetes Register, the Swedish Renal Registry, the Prescribed Drug Register, and the 2nd version of the Swedish-Danish Scandinavian Donations and Transfusions database. Cross-linking patient-level data is possible through the Personal Identity Number assigned to every individual who has resided in Sweden on a permanent basis. The Swedish Personal Identity Number is the unique identifier in all national registers.

Specifically, we aim:

1. To assess the importance of chronic kidney disease for prognosis after CABG.
2. To assess the consequences of acute kidney injury following CABG.
3. To analyze the prognosis in patients with depression prior to CABG.
4. To study risks and benefits of blood transfusions in cardiac surgery.
5. To study the risks associated with diabetes mellitus in cardiac surgery with special reference to type of diabetes (type 1 and type 2) and glycaemic control and duration of disease.
6. To investigate the long-term impact of different surgical strategies (e.g. use of multiple arterial grafts or non-use of cardio-pulmonary bypass) during CABG.
7. To analyze prognosis in relevant sub-populations undergoing CABG (e.g. patients 50 years or younger, possible differences between men and women, and patients with heart failure with preserved vs. reduced ejection fraction).
8. To investigate survival and morbidity in patients between 50 and 69 years undergoing aortic valve replacement with particular reference to prosthesis type (mechanical vs. biological).
9. To analyze the association between socioeconomic factors and prognosis in patients undergoing cardiac surgery.
10. To investigate factors related to durability of bioprosthetic aortic heart valves.

ELIGIBILITY:
Inclusion Criteria:

All adult patients who underwent cardiac surgery in Sweden during the study period

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who underwent cardiac surgery in Sweden during the study period
Sampling Method: Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2011-01; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 15 years

SECONDARY OUTCOMES:
Myocardial Infarction | 15 years
Heart Failure | 15 years
Stroke | 15 years
End-Stage Renal Disease | 15 years
Repeat Revascularization | 15 years
Cardiovascular Death | 15 years
Aortic valve reoperation | 15 years
Composite | 15 years
  Combined end-point of death and other secondary end-points

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Holzmann, MD, PhD, Principal Investigator — Karolinska Institutet, Karolinska University Hospital; Ulrik Sartipy, MD, PhD, Principal Investigator — Karolinska Institutet, Karolinska University Hospital

REFERENCES:
- [Derived] Dalen M, Persson M, Glaser N, Sartipy U. Socioeconomic Status and Risk of Bleeding After Mechanical Aortic Valve Replacement. J Am Coll Cardiol. 2022 Jun 28;79(25):2502-2513. doi: 10.1016/j.jacc.2022.04.030. PMID 35738711
- [Derived] Glaser N, Persson M, Franco-Cereceda A, Sartipy U. Cause of Death After Surgical Aortic Valve Replacement: SWEDEHEART Observational Study. J Am Heart Assoc. 2021 Nov 16;10(22):e022627. doi: 10.1161/JAHA.121.022627. Epub 2021 Nov 8. PMID 34743549
- [Derived] Dalen M, Nielsen S, Ivert T, Holzmann MJ, Sartipy U. Coronary Artery Bypass Grafting in Women 50 Years or Younger. J Am Heart Assoc. 2019 Sep 17;8(18):e013211. doi: 10.1161/JAHA.119.013211. Epub 2019 Sep 14. PMID 31522591
- [Derived] Glaser N, Persson M, Jackson V, Holzmann MJ, Franco-Cereceda A, Sartipy U. Loss in Life Expectancy After Surgical Aortic Valve Replacement: SWEDEHEART Study. J Am Coll Cardiol. 2019 Jul 9;74(1):26-33. doi: 10.1016/j.jacc.2019.04.053. PMID 31272548
- [Derived] Persson M, Edgren G, Dalen M, Glaser N, Olsson ML, Franco-Cereceda A, Holzmann MJ, Sartipy U. ABO blood type and risk of porcine bioprosthetic aortic valve degeneration: SWEDEHEART observational cohort study. BMJ Open. 2019 May 5;9(5):e029109. doi: 10.1136/bmjopen-2019-029109. PMID 31061061
- [Derived] Dalen M, Edgren G, Ivert T, Holzmann MJ, Sartipy U. Weekday and Survival After Cardiac Surgery-A Swedish Nationwide Cohort Study in 106 473 Patients. J Am Heart Assoc. 2017 May 16;6(5):e005908. doi: 10.1161/JAHA.117.005908. PMID 28512116
- [Derived] Glaser N, Jackson V, Holzmann MJ, Franco-Cereceda A, Sartipy U. Late Survival After Aortic Valve Replacement in Patients With Moderately Reduced Kidney Function. J Am Heart Assoc. 2016 Dec 17;5(12):e004287. doi: 10.1161/JAHA.116.004287. PMID 27988497
- [Derived] Glaser N, Jackson V, Holzmann MJ, Franco-Cereceda A, Sartipy U. Aortic valve replacement with mechanical vs. biological prostheses in patients aged 50-69 years. Eur Heart J. 2016 Sep 7;37(34):2658-67. doi: 10.1093/eurheartj/ehv580. Epub 2015 Nov 11. PMID 26559386
- [Derived] Sartipy U, Holzmann MJ, Hjalgrim H, Edgren G. Red Blood Cell Concentrate Storage and Survival After Cardiac Surgery. JAMA. 2015 Oct 20;314(15):1641-3. doi: 10.1001/jama.2015.8690. No abstract available. PMID 26501540
- [Derived] Dalen M, Ivert T, Holzmann MJ, Sartipy U. Household Disposable Income and Long-Term Survival After Cardiac Surgery: A Swedish Nationwide Cohort Study in 100,534 Patients. J Am Coll Cardiol. 2015 Oct 27;66(17):1888-97. doi: 10.1016/j.jacc.2015.08.036. PMID 26493661
- [Derived] Kuhl J, Sartipy U, Eliasson B, Nystrom T, Holzmann MJ. Relationship between preoperative hemoglobin A1c levels and long-term mortality after coronary artery bypass grafting in patients with type 2 diabetes mellitus. Int J Cardiol. 2016 Jan 1;202:291-6. doi: 10.1016/j.ijcard.2015.09.008. Epub 2015 Sep 12. PMID 26411993
- [Derived] Nystrom T, Holzmann MJ, Eliasson B, Kuhl J, Sartipy U. Glycemic Control in Type 1 Diabetes and Long-Term Risk of Cardiovascular Events or Death After Coronary Artery Bypass Grafting. J Am Coll Cardiol. 2015 Aug 4;66(5):535-43. doi: 10.1016/j.jacc.2015.05.054. PMID 26227192
- [Derived] Dalen M, Ivert T, Holzmann MJ, Sartipy U. Coronary artery bypass grafting in patients 50 years or younger: a Swedish nationwide cohort study. Circulation. 2015 May 19;131(20):1748-54. doi: 10.1161/CIRCULATIONAHA.114.014335. Epub 2015 Mar 18. PMID 25788458